CLINICAL TRIAL: NCT01896427
Title: Comparing Pain and Swelling After Surgical Extraction of Mandibular Third Molar in Dexamethasone Injection and Without Corticosteroid Methods
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohammad Javad Shirani (Other)
Collaborators: Isfahan University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Mohammad Javad Shirani, Dr, Isfahan University of Medical Sciences
Organization: Isfahan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 292037; 292037 (Other Grant/Funding Number: Isfahan University of Medical Sciences); IRCT2013042713140N1 (Registry Identifier: Iranian Registry of clinical trials)
Record Dates: First submitted 2013-06-30; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Oral Health; Molar, Third
Keywords: Third Molar; Edema; pain; trismus
MeSH Terms: conditions — Edema; Pain; Trismus | interventions — 21-benzyloxy-9alpha-fluoro-16alpha-methylpregna-1,4-dien-11beta,17alpha-diol-3,20-dione

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethazone IO (Active Comparator): For the case group, after the inferior alveolar block injection and before starting the surgery, single dose of dexamethasone (8mg) will injected into medial pterygoid and pterygomandibular space
  Interventions: Drug: 21-benzyloxy-9alpha-fluoro-16alpha-methylpregna-1,4-dien-11beta,17alpha-diol-3,20-dione
- Dexamethasone IM (Active Comparator): For the case group, after the inferior alveolar block injection and before starting the surgery, single dose of dexamethasone (8mg) will injected into medial pterygoid and pterygomandibular space
  Interventions: Drug: 21-benzyloxy-9alpha-fluoro-16alpha-methylpregna-1,4-dien-11beta,17alpha-diol-3,20-dione

INTERVENTIONS:
Drug: 21-benzyloxy-9alpha-fluoro-16alpha-methylpregna-1,4-dien-11beta,17alpha-diol-3,20-dione — single dose of dexamethasone (8mg) will injected

SUMMARY:
In some cases, impacted wisdom teeth should be extracted. Surgical extraction of these impacted third molars may provide special complication as pain, swelling, and trismus. In previous studies, some techniques as sutureless flap closure, modified flap designing, antibiotic usage, and injection of corticosteroids were presented. These methods are reducing post operative complications to moderate level. In this study, pain, swelling, trismus, general patients' satisfaction, and associated quality of life after the surgical removal of third mandibular impacted molars will be compared while injection of dexamethasone (8mg) does not need excessive time, effort, and equipments and it will be injected in numbness area into medial pterygoid muscle and pterygomandibular space to current corticosteroid injecting non-corticosteroid methods. To achieve this aim, 75 non pregnant participants have single impacted mandibular third molar in healthy and without pericoronitis manner, after provision of written informed consent will be entered to the study. During the study, unwilling participants to continue the study and those with abnormality of wound healing process will be excluded. The included participants will be assigned into three 25-people groups. The surgeries were done by 3 same instructed experienced oral and maxillofacial residents. After the surgery pain, swelling, trismus, general patients' satisfaction, and associated quality of life were evaluated using interview of questionnaire in 48 hour, 96 hour, and one week period of time. The comparison was done between these three groups.

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant participants have single impacted mandibular third molar in healthy and without pericoronitis manner
* They must have no contra-indication for injection of the corticosteroid and lidocaine with epinephrine
* Should not medicated by any possibly bias maker drug
* Type of the impaction, must not provide sever difficulty
* The participants should be mentally at healthy level and provide written informed consent to incorporate in the study

Exclusion Criteria:

-Unwilling participants to continue the study and those with abnormality of wound healing process

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain | 48 hours and one week after intervention
  Visual analogue scale of pain- Number of required analgesics tablets
Changes in Swelling | 48 hours and one week after intervention
  Questionnaire and VAS
Changes in Trismus | 48 hours and one week after intervention
  Questionnaire
Changes in General patients' satisfaction | 48 hours and one week after intervention
  Visual analogue scale for satisfaction
Changes in Quality of life | 96 hours and one week after intervention
  Questionnaire

SECONDARY OUTCOMES:
Trismus | one week period after the surgery
  Questionnaire about Maximum mouth opening- Patients complaint

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Movahedian, Oral and maxillofacial surgeon, Study Chair — Department of oral and maxillofacial surgery, Faculty of Dentistry, Isfahan University of Medical Sciences
Locations (1):
- Department of oral and maxillofacial surgery, Faculty of Dentistry, Isfahan University of Medical Sciences, Isfahan, Isfahan, Iran